CLINICAL TRIAL: NCT02843451
Title: Silymarin Treatment of Body Dysmorphic Disorder: A Double-Blind, Placebo-Controlled, Cross-Over Study
Brief Title: Milk Thistle in Body Dysmorphic Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Focus on other studies
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-0642
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Body Dysmorphic Disorder
MeSH Terms: conditions — Body Dysmorphic Disorders | interventions — milk-thistle extract; Silymarin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silymarin (Milk Thistle) (Experimental): Each subject will have a 4 week treatment phase with milk thistle.
  Interventions: Drug: Milk Thistle
- Placebo (Placebo Comparator): 4 week placebo phase before or after milk thistle phase depending on randomization.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Milk Thistle
  Other Names: Silymarin
  Arms: Silymarin (Milk Thistle)
Drug: Placebo
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The proposed study will consist of a 9 week double-blind cross-over study trial of milk thistle in 15 people (ages 18-65). The study will be divided into an initial 4 week phase, a one week wash out phase, and a second 4 week phase, with one of the 4 week phases consisting of active treatment with milk thistle, and the other 4 week phase consisting of inactive placebo treatment. Participants will be randomized to receive either milk thistle or placebo during the first 4 week phase on a 1:1 basis. This blinding will be maintained by the IDS pharmacy at the University of Chicago.

DETAILED DESCRIPTION:
The goal of the proposed study is to evaluate the efficacy and safety of silymarin (milk thistle) in adults with body dysmorphic disorder. The hypothesis to be tested is that silymarin will be more effective and well tolerated in adults with body dysmorphic disorder compared to placebo. The proposed study will provide needed data on the treatment of a disabling disorder that currently lacks a clearly effective treatment.

The primary aim of this application is to conduct a randomized placebo-controlled pharmacotherapy trial using silymarin (milk thistle) in 15 participants with body dysmorphic disorder. The study will consist of three phases: a 4 week active treatment phase with milk thistle, a 4 week placebo phase, and a one week wash out phase between the active and placebo phases. The subjects will be randomized to either receive active or placebo treatment in the first 4 weeks, and the other during the remaining 4 week phase.

This will be one of few studies assessing the use of pharmacotherapy for the treatment of body dysmorphic disorder in adults. Assessing the efficacy and safety of silymarin (milk thistle), will help inform clinicians about additional treatment options for adults suffering from this disorder.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18-65
* Diagnosis of current body dysmorphic disorder (BDD) based on DSM-5 criteria and confirmed using the clinician-administered Structural Clinical Interview for DSM-5 (SCID)
* Able and willing to provide written consent for participation

Exclusion Criteria:

* Unstable medical illness as determined by the investigator
* History of seizures
* Clinically significant suicidality (defined by the Columbia Suicide Severity Rating Scale)
* Baseline score greater than or equal to 17 on the Hamilton Depression Rating Scale (17-item HDRS)
* Lifetime history of bipolar disorder type I or II, schizophrenia, autism, any psychotic disorder, or any substance use disorder
* Initiation of psychotherapy of behavior therapy within 3 months prior to study baseline
* Previous treatment with milk thistle
* Any history of psychiatric hospitalization in the past year
* Currently pregnant (confirmed by urine pregnancy test)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale Modified for Body Dysmorphic Disorder (BDD-YBOCS) | Baseline and 9 weeks
  The entire study for the subject will last 9 weeks. Every four weeks and after the one week washout period the subject will take the BDD-YBOCS. The change in scores from baseline to after 9 weeks will be assessed. The scale itself assesses severity of body dysmorphic disorder symptoms.

SECONDARY OUTCOMES:
Clinical Global Impression- Severity and Improvement (CGI) | Baseline and 9 weeks
  The entire study for the subject will last 9 weeks. Every four weeks and after the one week washout period the subject will complete the CGI. The change in scores from baseline to after 9 weeks will be assessed. The scale itself assesses overall disorder severity.
Sheehan Disability Scale (SDS) | Baseline and 9 weeks
  The entire study for the subject will last 9 weeks. Every four weeks and after the one week washout period the subject will complete the SDS. The change in scores from baseline to after 9 weeks will be assessed. The scale itself assesses the level of disability from body dysmorphic disorder (or target disorder)
Hamilton Anxiety Rating Scale (HAM-A) | Baseline and 9 weeks
  The entire study for the subject will last 9 weeks. Every four weeks and after the one week washout period the subject will complete the HAM-A. The change in scores from baseline to after 9 weeks will be assessed. The scale itself assesses level of anxiety.
Hamilton Depression Rating Scale (HAM-D) | Baseline and 9 weeks
  The entire study for the subject will last 9 weeks. Every four weeks and after the one week washout period the subject will complete the HAM-D. The change in scores from baseline to after 9 weeks will be assessed. The scale itself assesses level of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, JD, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phillips KA, McElroy SL, Keck PE Jr, Pope HG Jr, Hudson JI. Body dysmorphic disorder: 30 cases of imagined ugliness. Am J Psychiatry. 1993 Feb;150(2):302-8. doi: 10.1176/ajp.150.2.302. PMID 8422082
- [Background] Buchanan BG, Rossell SL, Maller JJ, Toh WL, Brennan S, Castle DJ. Brain connectivity in body dysmorphic disorder compared with controls: a diffusion tensor imaging study. Psychol Med. 2013 Dec;43(12):2513-21. doi: 10.1017/S0033291713000421. Epub 2013 Mar 11. PMID 23473554
- [Background] Dunai J, Labuschagne I, Castle DJ, Kyrios M, Rossell SL. Executive function in body dysmorphic disorder. Psychol Med. 2010 Sep;40(9):1541-8. doi: 10.1017/S003329170999198X. Epub 2009 Dec 2. PMID 19951448
- [Background] Phillips KA, Albertini RS, Rasmussen SA. A randomized placebo-controlled trial of fluoxetine in body dysmorphic disorder. Arch Gen Psychiatry. 2002 Apr;59(4):381-8. doi: 10.1001/archpsyc.59.4.381. PMID 11926939
- [Background] Phillips KA. Pharmacologic treatment of body dysmorphic disorder: review of the evidence and a recommended treatment approach. CNS Spectr. 2002 Jun;7(6):453-60, 463. doi: 10.1017/s109285290001796x. PMID 15107767
- [Background] Yaghmaei P, Oryan S, Mohammadi K, Solati J. Role of serotonergic system on modulation of depressogenic-like effects of silymarine. Iran J Pharm Res. 2012 Winter;11(1):331-7. PMID 24250456
- [Background] Lu P, Mamiya T, Lu L, Mouri A, Niwa M, Kim HC, Zou LB, Nagai T, Yamada K, Ikejima T, Nabeshima T. Silibinin attenuates cognitive deficits and decreases of dopamine and serotonin induced by repeated methamphetamine treatment. Behav Brain Res. 2010 Mar 5;207(2):387-93. doi: 10.1016/j.bbr.2009.10.024. Epub 2009 Oct 24. PMID 19857526
- [Background] Seamans JK, Yang CR. The principal features and mechanisms of dopamine modulation in the prefrontal cortex. Prog Neurobiol. 2004 Sep;74(1):1-58. doi: 10.1016/j.pneurobio.2004.05.006. PMID 15381316
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Phillips KA, Hollander E, Rasmussen SA, Aronowitz BR, DeCaria C, Goodman WK. A severity rating scale for body dysmorphic disorder: development, reliability, and validity of a modified version of the Yale-Brown Obsessive Compulsive Scale. Psychopharmacol Bull. 1997;33(1):17-22. PMID 9133747
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] Burker EJ, Evon DM, Marroquin Loiselle M, Finkel JB, Mill MR. Coping predicts depression and disability in heart transplant candidates. J Psychosom Res. 2005 Oct;59(4):215-22. doi: 10.1016/j.jpsychores.2005.06.055. PMID 16223624